CLINICAL TRIAL: NCT06795737
Title: Effectiveness and Safety of Exercise-based Cardiac Rehabilitation (ExCR) During the Vulnerable Period in Patients With Acute Decompensated Heart Failure (ADHF): A Randomized Controlled Trial
Brief Title: ExCR's Effects and Safety in Vulnerable ADHF Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YE Jing (Other)
Responsible Party: Sponsor-Investigator, YE Jing, Chief Nurse of the Cardiovascular Intensive Care Unit, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Peaking UFH
Record Dates: First submitted 2024-12-19; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
Keywords: Acute Decompensated Heart Failure (ADHF)；Vulnerable Phase；Exercise Rehabilitation；RCT
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Exercise rehabilitation
  Interventions: Behavioral: Exercise rehabilitation
- Control group (Sham Comparator): Conventional rehabilitation
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Exercise rehabilitation — The experimental group's protocol consists of two stages: in-hospital Phase I and post-discharge self-training. For Phase I, cardiac and rehab specialists assess NYHA classification, muscle strength, and mobility to create an exercise plan, supervised by therapists and nurses. Phase II involves twice-weekly outpatient rehab for 24 sessions and weekly remote guidance with WeChat and wristbands to track vitals, totaling 12 remote sessions. Exercise prescriptions are customized based on 6MWTD outcomes, with ongoing support from rehab staff and nurses.
  Arms: Experimental group
Behavioral: Conventional rehabilitation — Health Education: Nurses provide manuals on heart failure causes, treatment, diet, exercise (detailing frequency, intensity, duration, types, and safety), and self-monitoring to control group patients.
  Outpatient Follow-up: Post-discharge, heart failure patients have follow-ups at 2 weeks, 1 month, 2 months, and 3 months. A multidisciplinary team of doctors, pharmacists, and nurses handles these, with doctors for assessment, pharmacists for medication education, and nurses for self-care assessment and education.
  Arms: Control group

SUMMARY:
Exercise-based cardiac rehabilitation has become a key component of the comprehensive care system for patients with stable heart failure (HF). However, due to hemodynamic instability and functional decline in early ADHF, most HF rehab studies exclude current/recent ADHF exacerbations. Currently, ADHF management strategies lack robust evidence, and the timing, duration, and frequency of exercise interventions need further validation globally.

This study aims to address the following issues:

Develop an exercise management program for ADHF patients, verify its feasibility, and determine the safety and applicability of early exercise rehabilitation; Evaluate the improvement of participants in terms of physical function, cardiac function, and quality of life.

The research team will compare the formulated exercise rehabilitation program with conventional rehabilitation guidance to verify its feasibility and effectiveness.

Participants will:

Physicians and rehabilitation therapists will comprehensively assess the participants' conditions to determine the start time of rehabilitation training. Based on the patients' cardiac function, muscle strength, and heart failure-related clinical indicators, rehabilitation training is divided into two stages (the first stage is early in-hospital training, and the second stage is self-directed training after discharge). Exercise types mainly include respiratory training, bed activities, rehabilitation pedaling, and resistance training. Rehabilitation therapists and nurses will monitor participants' vital signs during the exercise process and choose the appropriate exercise intensity based on the participants' level of fatigue.

The exercise rehabilitation program will be evaluated and adjusted every two weeks for a total period of 12 weeks.

At the time of enrollment, discharge, two weeks after discharge, and four weeks after discharge, participants will need to complete questionnaires, including demographic and disease condition surveys, grip strength tests, Activities of Daily Living (ADL) scales, Short Physical Performance Battery (SPPB) scales, Minnesota Living with Heart Failure Questionnaire (MLHFQ) scales, and 6-minute walk tests, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized for ADHF for over 24 hours.
2. Age 18-80 years.
3. At least one acute heart failure symptom: dyspnea at rest or exertion, fatigue, orthopnea, or paroxysmal nocturnal dyspnea.
4. At least two heart failure signs: confirmed pulmonary congestion or edema on exam or chest X-ray, jugular venous distension, peripheral edema, rapid weight gain (>2 kg in 3 days), or elevated BNP (≥100 ng/L) and NT-proBNP (≥300 ng/L).
5. Change in heart failure treatment plan with initiation or increased dosage of: diuretics, vasodilators, positive inotropic agents (e.g., digoxin), or other neurohormonal modulators (ACEI/ARB/ARNI, β-blocker, MRA).

Exclusion Criteria:

1. Indications for urgent cardiovascular surgery (e.g., heart transplantation, left ventricular assist device).
2. Cardiogenic shock.
3. Recent deep vein thrombosis.
4. Severe cardiovascular diseases (e.g., severe aortic stenosis, mitral regurgitation).
5. GFR <30 ml/min or need for dialysis during the study.
6. Severe COPD (FEV1/FVC <0.7 post-bronchodilator, with severe defined as 30% ≤ FEV1 <50% predicted, and very severe as FEV1 <30% predicted).
7. Severe frailty (Clinical Frailty Scale CFS ≥7).
8. Mental, psychological, cognitive disorders, or substance dependence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the 6-minute walking test distance | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Assess the changes in participants' 6MWT distance at baseline and 1, 2, and 3 months post-discharge.

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction （LVEF%） | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Assess the changes in participants' LVEF% at baseline and 1, 2, and 3 months post-discharge.
Brain Natriuretic Peptide（BNP） | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Assess the changes in participants' BNP at baseline and 1, 2, and 3 months post-discharge.
NYHA class | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Assess the changes in participants' NYHA class at baseline and 1, 2, and 3 months post-discharge.
Grip strength | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Assess grip strength using a dynamometer（CAMRY brand electronic hand dynamometer）; participants squeeze twice with their dominant hand and record the average.
Length of hospitalization | From hospitalization to discharge, an average of 12 weeks.
  Length of hospitalization will be compared between intervention and control groups at discharge.
Short Physical Performance Battery（SPPB） | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  SPPB : Assesses physical performance with three tests: balance, 4-meter gait speed, and repeated chair stands. Each test scores 0-4; total score 0-12. Scores: 0-6 (poor), 7-9 (moderate), 10-12 (good).The SPPB scale will assess participants' physical performance at enrollment and 1, 2, and 3 months post-discharge.
Activities of Daily Living（ADL） | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Barthel Index: 10 items (feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, transfers, walking, stairs). Each item scored 0, 5, 10, 15; total 0-100. ≤40: severe dependence; 41-60: moderate; 61-99: mild; 100: independent. Higher scores indicate greater self-care ability.The Barthel Index will be used to assess ADL changes in participants at baseline and 1, 2, and 3 months post-discharge.
Quality of life using MLHFQ scale | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  MLHFQ scale: 21-item questionnaire assessing heart failure's impact on quality of life over the past month. Three domains: physical (8 items), emotional (5 items), and other (8 items). Each item scored 0-5 (0=none, 1=rarely, 2=occasionally, 3=sometimes, 4=often, 5=always). Total score: 0-105. Higher scores indicate worse quality of life; lower scores indicate better quality of life.The Minnesota Living with Heart Failure Questionnaire will be used to assess QoL changes in participants at baseline and 1, 2, and 3 months post-discharge.
Degree of frailty. | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Clinical Frailty Scale: 1-9 scale (very fit, well, managing well, vulnerable, mildly frail, moderately frail, severely frail, very severely frail, terminally ill). Score ≥5 indicates frailty.The Clinical Frailty Scale will be used to assess frailty changes in participants at baseline and at 1, 2, and 3 months post-discharge.

OTHER OUTCOMES:
3-month all-cause readmission rate | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  The 3-month all-cause readmission rate of study participants post-discharge.Assessment at 3 months post-discharge.
3-month all-cause mortality rate | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  The 3-month all-cause mortality rate of study participants post-discharge.Assessment at 3 months post-discharge.
Adverse events | From enrollment to the end of the 12-week exercise rehabilitation intervention.
  Adverse events will be monitored and recorded throughout the study. Data will be collected on falls, injuries, musculoskeletal issues, major cardiovascular events, and any other events potentially related to study protocol implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ye, MSN., Study Chair — Peaking University First Hospital; Yimeng Jiang, Ph.D., Study Director — Peaking University First Hospital; Lihua Zhao, MSN., Principal Investigator — Peaking University First Hospital; Wenhui Ding, Prof., Principal Investigator — Peaking University First Hospital; Xiaoning Han, Ph.D., Principal Investigator — Peaking University First Hospital; Lei Yang, Principal Investigator — Peaking University First Hospital; Yuling Wang, Principal Investigator — Peaking University First Hospital; Baiyu Zhang, Principal Investigator — Peaking University First Hospital; Zhuo Zhao, Principal Investigator — Peaking University First Hospital
Locations (1):
- Peaking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chioncel O, Mebazaa A, Maggioni AP, Harjola VP, Rosano G, Laroche C, Piepoli MF, Crespo-Leiro MG, Lainscak M, Ponikowski P, Filippatos G, Ruschitzka F, Seferovic P, Coats AJS, Lund LH; ESC-EORP-HFA Heart Failure Long-Term Registry Investigators. Acute heart failure congestion and perfusion status - impact of the clinical classification on in-hospital and long-term outcomes; insights from the ESC-EORP-HFA Heart Failure Long-Term Registry. Eur J Heart Fail. 2019 Nov;21(11):1338-1352. doi: 10.1002/ejhf.1492. Epub 2019 May 24. PMID 31127678
- [Background] Pack QR, Priya A, Lagu T, Pekow PS, Berry R, Atreya AR, Ades PA, Lindenauer PK. Cardiac Rehabilitation Utilization During an Acute Cardiac Hospitalization: A NATIONAL SAMPLE. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):19-26. doi: 10.1097/HCR.0000000000000374. PMID 30586111
- [Background] Patti A, Merlo L, Ambrosetti M, Sarto P. Exercise-Based Cardiac Rehabilitation Programs in Heart Failure Patients. Heart Fail Clin. 2021 Apr;17(2):263-271. doi: 10.1016/j.hfc.2021.01.007. Epub 2021 Feb 12. PMID 33673950
- [Background] Lesyuk W, Kriza C, Kolominsky-Rabas P. Cost-of-illness studies in heart failure: a systematic review 2004-2016. BMC Cardiovasc Disord. 2018 May 2;18(1):74. doi: 10.1186/s12872-018-0815-3. PMID 29716540
- [Background] Taylor RS, Walker S, Smart NA, Piepoli MF, Warren FC, Ciani O, Whellan D, O'Connor C, Keteyian SJ, Coats A, Davos CH, Dalal HM, Dracup K, Evangelista LS, Jolly K, Myers J, Nilsson BB, Passino C, Witham MD, Yeh GY; ExTraMATCH II Collaboration. Impact of Exercise Rehabilitation on Exercise Capacity and Quality-of-Life in Heart Failure: Individual Participant Meta-Analysis. J Am Coll Cardiol. 2019 Apr 2;73(12):1430-1443. doi: 10.1016/j.jacc.2018.12.072. PMID 30922474
- [Background] Maddocks S, Cobbing S. Patients' Experiences of and Perspectives on Phase 1 Cardiac Rehabilitation after Coronary Artery Bypass Graft Surgery. Physiother Can. 2017;69(4):333-340. doi: 10.3138/ptc.2016-39GH. PMID 30369701
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Zou CH, Zhang J. [Interpretation of 2023 ESC focused update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure]. Zhonghua Xin Xue Guan Bing Za Zhi. 2023 Dec 24;51(12):1268-1272. doi: 10.3760/cma.j.cn112148-20230908-00143. Chinese. PMID 38123211
- [Derived] Ye J, Zhao L, Jiang Y, Hu L, Yang L, Wang Y, Ding W, Zheng Y. Effectiveness and safety of exercise-based cardiac rehabilitation (ExCR) during the vulnerable period in patients with acute decompensated heart failure (ADHF): a randomised controlled trial protocol. BMJ Open. 2025 Sep 21;15(9):e102812. doi: 10.1136/bmjopen-2025-102812. PMID 40976670